CLINICAL TRIAL: NCT04548297
Title: Clinical Factors Associated With Position Sense in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cagla Ozkul, Research Assistant, Gazi University
Other Study IDs: 2020-122
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; sensation; fatigue; physical activity
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Motor Activity | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Multiple Sclerosis: MS patients (EDSS: 0-5,5)
  Interventions: Other: Assessment
- Healthy group: Healthy individuals without chronic disease
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Assessments of foot sole sensation, joint position sensation, attention, fatigue, body awareness, and physical activity level

SUMMARY:
Sensory impairment is an important problem for patients with Multiple Sclerosis (MS). Although there is no complete loss of sensation in patients, 80% of patients have a significant sensory impairment. The sensory system plays an important role in providing the feedback required to perform motor tasks. Cutaneous sensation, especially in the sole of the foot, is very important in maintaining balance and gait. There are studies showing decreased foot sole sensation in MS patients. Another sensation that is important during motor tasks is the proprioceptive sensation.

The aim of this study is to examine the relationship between the sensation of foot sole and joint position, clinical features, attention, fatigue, body awareness and physical activity level in patients with MS.

DETAILED DESCRIPTION:
Patients with MS between 0-5,5 score according to the Extended Disability Status Scale (EDSS) and healthy individuals of similar age and sex to patients will be included in the study. The sensation of foot sole, joint position sensation, attention, fatigue, body awareness, and physical activity level will be evaluated.

The investigators will use t-tests to compare for quantitative variables and chi-square for the categorical variables between groups. In addition, the investigators will examine the correlations between the sensation of the foot sole, joint position sensation, attention, fatigue, body awareness, and physical activity level using Pearson bivariate correlations.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Having a diagnosis of "Multiple Sclerosis"
* Relapse free in the last 3 mounts
* Ambulatory status (Expanded Disability Status Scale score ≤ 6 )
* No diagnosis of depression

Exclusion Criteria:

* Any cardiovascular, orthopedic, visual, and hearing problems that may affect the results of the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ambulatory sample
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Light touch-pressure sensation | 10 minutes
  Light touch-pressure sensation will be assessed using a full Semmes-Weinstein Monofilament (SWM) test kit (North Coast Medical, San Jose, CA, USA).
Vibration sensation | 10 minutes]
  Duration of vibration sensation will be measured using 128-Hz frequency tuning fork (Elcon1 Medical Instruments, Tuttlingen, Germany).
position sensation of knee joint | 5 minutes
  Open kinetic chain position of both knees will be evaluated using a Dualer IQ Digital Inclinometer (J-Tech Medical, Midvale, UT, USA).
Knee proprioception | 10 minutes
  Knee proprioception will be evaluated with the active joint reposition test using the isokinetic system (Cybex Norm, Humac, CA, USA).

SECONDARY OUTCOMES:
Fatigue Severity | 5 minutes
  In the Fatigue Severity Scale (FSS), participants are asked to rate their fatigue level between 1 and 7 in the 9 statements (including motivation, exercise, physical functioning, carrying out duties, and interfering with work, family, or social life) during the last week.The minimum score possible is 9 and the highest is 63. The higher score indicates more severe fatigue.
attention | 5 minutes
  Attention will be evaluated by Trail Making Test.
Physical Activity | 10 minutes
  Physical Activity will be evaluated using International Physical Activity Questionnaires (IPAQ). The IPAQ measures vigorous-intensity activity, moderate-intensity activity, and walking activity levels by calculating physically active time in regard to the number of days and average time per day in the last week. The activity levels are represented as a Metabolic Equivalent of Tasks (METs) which is the energy expended during sitting at rest. The total score of IPAQ indicates a low physical activity of fewer than 600 MET-minutes per week, moderate physical activity of more than 600 MET-minutes per week, and a high level of physical activity of more than 3000 MET-minutes per week. The higher score indicates a greater physical activity level of the person.
Body Awareness | 5 minutes
  The Body Awareness Questionnaire is an 18-item scale designed to assess self-reported attentiveness to normal non-emotive body processes, specifically, sensitivity to body cycles and rhythms, ability to detect small changes in normal functioning, and ability to anticipate bodily reactions. Each item is rated ranging from 1 (totally agree) to 7 (totally disagree). The minimum score possible is 18 and the highest is 126. The higher score indicates more awareness of the body.

CONTACTS AND LOCATIONS:
Overall Officials: Cagla Ozkul, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sanders EA, Arts RJ. Paraesthesiae in multiple sclerosis. J Neurol Sci. 1986 Jul;74(2-3):297-305. doi: 10.1016/0022-510x(86)90115-2. PMID 3734839
- [Background] Merchut MP, Gruener G. Quantitative sensory threshold testing in patients with multiple sclerosis. Electromyogr Clin Neurophysiol. 1993 Mar;33(2):119-24. PMID 8449168
- [Background] Kars HJ, Hijmans JM, Geertzen JH, Zijlstra W. The effect of reduced somatosensation on standing balance: a systematic review. J Diabetes Sci Technol. 2009 Jul 1;3(4):931-43. doi: 10.1177/193229680900300441. PMID 20144343
- [Background] Eils E, Behrens S, Mers O, Thorwesten L, Volker K, Rosenbaum D. Reduced plantar sensation causes a cautious walking pattern. Gait Posture. 2004 Aug;20(1):54-60. doi: 10.1016/S0966-6362(03)00095-X. PMID 15196521
- [Derived] Eldemir K, Ozkul C, Yildirim MS, Eldemir S, Saygili F, Irkec C, Guclu-Gunduz A. Relationship between lower extremity sensation, physical activity, cognition, body awareness, and fatigue in people with multiple sclerosis: a cross-sectional study. Acta Neurol Belg. 2025 Jun;125(3):801-810. doi: 10.1007/s13760-025-02768-1. Epub 2025 Mar 26. PMID 40133734